CLINICAL TRIAL: NCT02105974
Title: A 12-Week Study to Evaluate the Efficacy and Safety of Fluticasone Furoate/Vilanterol Inhalation Powder (FF/VI) 100/25 mcg Once Daily Compared With Vilanterol Inhalation Powder (VI) 25 mcg Once Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study Evaluating the Efficacy and Safety of Fluticasone Furoate/Vilanterol Inhalation Powder (FF/VI) Compared With Vilanterol Inhalation Powder (VI) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200820
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Fluticasone Furoate (FF); Vilanterol (VI); Dry Powder Inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/Vilanterol 100/25 Inhalation Powder (Experimental): Inhaled corticosteroid (ICS)/long-acting beta2-agonist (LABA)
  Interventions: Drug: Fluticasone Furoate/Vilanterol
- Vilanterol 25 Inhalation Powder (Experimental): Long-acting beta2-agonist (LABA)
  Interventions: Drug: Vilanterol

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol — 100 mcg FF micronized drug blended with lactose per blister in one strip and 25 mcg VI micronized drug blended with lactose and magnesium stearate per blister in another strip, administered together by ELLIPTA™ inhaler
  Arms: Fluticasone Furoate/Vilanterol 100/25 Inhalation Powder
Drug: Vilanterol — 25 mcg of Vilanterol micronized drug (as the 'M' salt triphenylacetate) blended with lactose and magnesium stearate per blister in one strip and lactose in another strip, administered together by ELLIPTA™ inhaler
  Arms: Vilanterol 25 Inhalation Powder

SUMMARY:
This is a Phase IIIa, multicenter, randomized, stratified (reversibility status), double-blind, parallel-group study to evaluate the efficacy and safety of FF/VI 100/25 micrograms (mcg) once daily (QD) compared with VI 25 mcg QD, administered in the morning via the ELLIPTA™ inhaler. The primary objective of this study is to evaluate the contribution on lung function (as measured by trough forced expiratory volume in one second [FEV1]) of FF 100 mcg to the FF/VI 100/25 mcg QD combination by comparison of the latter with VI 25 mcg QD and the safety of FF/VI 100/25 mcg over a 12-week treatment period in subjects with COPD. ELLIPTA™ is a registered trademark of GlaxoSmithKline.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed consent: Subjects must give their signed and dated written informed consent to participate
* Gender: Male subjects or female subjects. Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy. The decision to include or exclude women of childbearing potential may be made at the discretion of the investigator in accordance with local practice in relation to adequate contraception.
* Age: >=40 years of age at Screening (Visit 1)
* COPD diagnosis: Subjects with a clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society: COPD is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it is also associated with significant systemic consequences.
* Severity of disease: Subjects with a measured post-albuterol (salbutamol) FEV1/ Forced Vital Capacity (FVC) ratio of <=0.70 and FEV1 >=30 to <=70 percent of predicted normal values using Global Lung Function Initiative 2012 reference equations at Screening (Visit 1).
* Tobacco use: Subjects with a current or prior history of >=10 pack-years of cigarette smoking at Screening (Visit 1). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* History of COPD exacerbation: A documented history (e.g., medical record verification) of at least one COPD exacerbation in the 12 months prior to Screening (Visit 1) that required either systemic/oral corticosteroids, antibiotics and/or hospitalization.
* Current symptoms of COPD: A Subject Diary combined symptom score (combination of breathlessness, cough, sputum, and night time awakenings requiring treatment with albuterol [salbutamol]) of >=4 on at least 5 of the 7 days immediately preceding Visit 2 (Randomization)
* QTc Criteria: QTc <450 msec or QTc <480 msec for patients with bundle branch block.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Other respiratory disorders: Subjects with alpha1-antitrypsin deficiency as the underlying cause of COPD as the underlying cause of COPD, active tuberculosis, lung cancer, bronchiectasis (Note: focal bronchiectasis is not exclusionary), sarcoidosis, pulmonary fibrosis (Note: focal fibrotic pulmonary lesions are not exclusionary), primary pulmonary hypertension, interstitial lung diseases, or other active pulmonary diseases.
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* Chest X-ray (or computed tomography [CT] scan): Subjects with a chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Screening (Visit 1) if a chest X-ray or CT scan is not available within 1 year prior to Screening (Visit 1).
* Hospitalization: Subjects who are hospitalized due to poorly controlled COPD that has not resolved at least 4 weeks prior to Screening (Visit 1) and at least 6 weeks following the last dose of systemic corticosteroids.
* Poorly controlled COPD: Subjects with poorly controlled COPD, defined as the occurrence of any of the following in the 6 weeks prior to Screening (Visit 1): Acute worsening of COPD that is managed by subject with systemic corticosteroids or antibiotics or that requires treatment prescribed by a physician.
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Screening (Visit 1).
* COPD exacerbation/lower respiratory tract infection during the Run-In Period: Subjects who experience a moderate/severe COPD exacerbation (As per definition of "COPD Exacerbations and Pneumonia" in protocol) and/or a lower respiratory tract infection (including pneumonia) during the Run-In Period.
* Abnormal, clinically significant laboratory finding: Subjects who have an abnormal clinical significant finding in any liver chemistry test at Screening (Visit 1) or upon repeat prior to randomization.
* Abnormal, clinically significant 12-lead ECG at Screening (Visit 1): Subjects who have an abnormal, clinically significant 12-Lead electrocardiogram (ECG) finding at Screening (Visit 1) or upon repeat prior to randomization.
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant and unstable disease such as cardiovascular (e.g., patients requiring implantable cardioverter-defibrillators (ICD), pacemaker requiring a rate set >60 beats per minute (bpm), uncontrolled hypertension, New Your Heart Association Class IV, known left ventricular ejection fraction <30 percent) neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), peptic ulcer disease, or hematological abnormalities.
* Liver disease: Subjects who have unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Subjects with chronic stable hepatitis B and C are eligible if the subject otherwise meets entry criteria (e.g., presence of hepatitis B surface antigen or positive hepatitis C test result within 3 months of screening). However, subjects with chronic stable hepatitis B are excluded if significant immunosuppressive or cytotoxic agents are administered, due to risk of hepatitis B reactivation, unless the hepatitis B antivirals are administered as outlined in the Chronic Hepatitis B American Association for the Study of Liver Diseases' (AASLD) Practice Guidelines.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Contraindications: Subjects with a history of allergy or hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroids) or components of the inhalation powder (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the investigator, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol (salbutamol) or their ipratropium bromide for the 4-hour period required prior to spirometry testing at each study visit.
* Additional medication: Use of certain medications such as bronchodilators and corticosteroids for the protocol-specific times prior to Visit 1 (the Investigator will discuss the specific medications)"
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen as needed (prn) use (i.e., <=12 hours per day) is not exclusionary.
* Sleep apnea: Subjects with clinically significant sleep apnea who require use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV).
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening (Visit 1) or who will enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded.
* Non-Compliance during Run-In Period: Failure to demonstrate adequate compliance defined as completion of Diary Card (completed all diary entries on at least 5 of the last 7 consecutive days), the ability to withhold anti-COPD medications and to keep clinic visit appointments. In addition, subjects must have recorded the Run-In study medication use on at least 5 of the last 7, consecutive days of the Run-In period to continue in the study.
* Potential of non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Prior use of study medication/other investigational drugs: Subjects who have received an investigational drug within 30 days of entry into this study (Screening), or within 5 drug half-lives of the investigational drug, whichever is longer. Note: Subjects who participated in a previously completed study and/or were excluded/ withdrawn from an ongoing study that included/includes FF/VI and/or VI are eligible to participate in the current study, if they have not received investigational study medication within 30 days of Screening (Visit 1).
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1621 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2015-07-08 (Actual); Study Completion 2015-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (120):
- United States (17):
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Morgantown, West Virginia
- Bulgaria (7):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Vidin
- Germany (15):
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Japan (30):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Yamaguchi
- Poland (7):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Romania (9):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Suceava
- Russia (8):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Khantymansiysk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
- South Africa (11):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Welkom, Free State
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Tygerberg
- South Korea (5):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Taiwan (3):
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Taichung
- Ukraine (8):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kremenchuk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Siler TM, Nagai A, Scott-Wilson CA, Midwinter DA, Crim C. A randomised, phase III trial of once-daily fluticasone furoate/vilanterol 100/25 mug versus once-daily vilanterol 25 mug to evaluate the contribution on lung function of fluticasone furoate in the combination in patients with COPD. Respir Med. 2017 Feb;123:8-17. doi: 10.1016/j.rmed.2016.12.001. Epub 2016 Dec 2. PMID 28137501
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200820 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Par meeting continuation criteria during the run-in period were randomized (1:1) to receive fluticasone furoate (FF)/vilanterol (VI) or VI. Of the 2423 par screened, 1622 were randomized. 1620 received at least one dose of double-blind study medication and comprised the Intent-to-Treat population.
Pre-assignment Details: Participants(par) with a history of chronic obstructive pulmonary disease(COPD) meeting eligibility criteria at screening were enrolled in a 2-week, single-blind(placebo) run-in period to obtain baseline use of albuterol(salbutamol), COPD symptom scores and disease stability.
Groups:
- Placebo Run-In: Participants received placebo once daily (QD) in the morning for 2 weeks. In addition, participants were provided an inhaled short-acting beta2-receptor agonist (SABA), albuterol (salbutamol) (metered dose inhaler [MDI] or nebules), to be used as a rescue medication for relief of chronic obstructive pulmonary disease (COPD) symptoms during the Run-in and Treatment Periods.
- FF/VI 100/25 µg QD: Participants received fluticasone furoate/vilaterol (FF/VI) 100/25 microgram(µg) inhalation via a dry powder inhaler (DPI) once daily (QD) in the morning for 12 weeks. In addition, all participants were provided with albuterol (salbutamol) or oxitropium bromide (applicable sites in Japan) to be used as rescue medication (via metered-dose inhaler [MDI] or nebules) for relief of COPD symptoms during the Run-In and Treatment Periods.
- VI 25 µg QD: Participants received VI 25 µg inhalation QD via a DPI in the morning for 12 weeks. In addition, all participants were provided with albuterol (salbutamol) or oxitropium bromide (applicable sites in Japan) to be used as rescue medication (via metered-dose inhaler [MDI] or nebules) for relief of COPD symptoms during the Run-In and Treatment Periods.
Period: 2 Week Run-in Period
Arm/Group | Placebo Run-In | FF/VI 100/25 µg QD | VI 25 µg QD
Started | 2423 | 0 | 0
Completed | 1622 | 0 | 0
Not Completed | 801 | 0 | 0
Not completed — Withdrew during pre-screen period | 158 | 0 | 0
Not completed — Did not meet inclusion/exclusion criteri | 603 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0
Not completed — Study closed/terminated | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrew consent | 23 | 0 | 0
Not completed — Investigator discretion | 8 | 0 | 0
Period: 12 Week (Wk) Treatment Period (TP)
Arm/Group | Placebo Run-In | FF/VI 100/25 µg QD | VI 25 µg QD
Started | 0 | 806 | 814
Completed the Treatment(Trt) Period | 0 | 764 (Par completed TP if attended Visit (V7, Wk12), did not withdraw at V7 and did not stop trt before V7) | 754 (Par completed TP if attended Visit (V7, Wk12), did not withdraw at V7 and did not stop trt before V7)
Completed | 0 | 764 (Par. completed study if attended visit 7, had follow-up contact and no early withdrawal) | 756 (Par. completed study if attended visit 7, had follow-up contact and no early withdrawal)
Not Completed | 0 | 42 | 58
Not completed — Adverse Event | 0 | 14 | 18
Not completed — Lack of Efficacy | 0 | 6 | 9
Not completed — Protocol deviation | 0 | 2 | 6
Not completed — Participant reached stopping criteria | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 7 | 4
Not completed — Withdrawal by Subject | 0 | 12 | 18

BASELINE CHARACTERISTICS:
Groups:
- FF/VI 100/25 µg QD: Participants received fluticasone furoate/vilaterol (FF/VI) 100/25 microgram(µg) inhalation via a dry powder inhaler (DPI) once daily (QD) in the morning for 12 weeks. In addition, all participants were provided with albuterol (salbutamol) or oxitropium bromide (applicable sites in Japan) to be used as rescue medication (via metered-dose inhaler (MDI) or nebules) for relief of COPD symptoms during the Run-In and Treatment Periods.
- VI 25 µg QD: Participants received VI 25 µg inhalation QD via a DPI in the morning for 12 weeks. In addition, all participants were provided with albuterol (salbutamol) or oxitropium bromide (applicable sites in Japan) to be used as rescue medication (via metered-dose inhaler (MDI) or nebules) for relief of COPD symptoms during the Run-In and Treatment Periods.
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg QD | VI 25 µg QD | Total
Number analyzed (Participants) | 806 | 814 | 1620
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (8.58) | 65.4 (9.02) | 65.3 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 189 | 390
  Male | 605 | 625 | 1230
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6 | 10 | 16
  Asian - East Asian Heritage | 77 | 77 | 154
  Asian - Japanese Heritage | 185 | 185 | 370
  White - White/Caucasian/European Heritage | 538 | 541 | 1079
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (BL) in Clinic Visit Trough (Pre-bronchodilator and Pre-dose) FEV1, on Treatment Day 84
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 14, 28, 56 and 84. BL was defined as the mean of the assessments made 30 minutes pre-dose and immediately pre-dose on Treatment Day 1.Trough FEV1 was defined as the mean of the FEV1 values obtained 23 and 24 hours after previous morning's dosing. Change from BL was calculated as the average at each visit minus the BL value. Analysis was performed using a repeated measures model with covariates of treatment, reversibility status (stratum), BL, region, day, day by BL and day by treatment interactions.
Time Frame: Baseline to Day 84
Population: Intent-to-Treat (ITT) Population: all randomized par. who received at least one dose of study medication. Number of par. presented represent those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | FF/VI 100/25 µg QD | VI 25 µg QD
Number analyzed (Participants) | 759 | 749
Liter | 0.116 (0.0074) | 0.082 (0.0075)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD vs VI 25 µg QD; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least Squares Mean Difference = 0.034, 95% CI 2-sided [0.014 to 0.055]

2. Secondary Outcome: Percentage of Rescue-free 24-hour Periods Over the Entire 12-week Treatment Period
Description: Participants were given daily record cards for daily completion from BL (Week -1) through Week 12 (Visit 7) each morning and prior prior to taking study medication (i.e., single-blind and double-blind study medication), supplemental medication (albuterol [salbutamol] if received). Participants recorded number of occasions supplemental albuterol/salbutamol (MDI and/or nebules) or oxitropium bromide (applicable sites in Japan) used over the previous 24 hours and any medical problems that they had experienced and any medication used to treat these medical problems over the previous 24 hours. Rescue-free 24-hour periods are defined as the 24-hour periods in which the rescue medication (albuterol [salbutamol]) was not used. The percentage of 24-hour periods are summarized for the entire treatment period (12 weeks). Analysis was performed using an analysis of covariance (ANCOVA) model with covariates of treatment, reversibility status (stratum), baseline (week -1) and region.
Time Frame: BL (Week -1), Week 1 to Week 12
Population: ITT Population, all randomized participants who received at least one dose of study medication. Only those participants with at least 1 on treatment rescue medication measurement during the treatment period and without missing covariate information were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free periods
Arm/Group | FF/VI 100/25 µg QD | VI 25 µg QD
Number analyzed (Participants) | 801 | 802
Percentage of rescue-free periods | 47.03 (1.070) | 44.41 (1.069)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD vs VI 25 µg QD; Test type: Superiority or Other; p = 0.084, ANCOVA; Least Squares Mean Difference = 2.62, 95% CI 2-sided [-0.35 to 5.59]

3. Secondary Outcome: Time to First On-treatment Occurrence of Moderate or Severe COPD Exacerbation
Description: Time to first on-treatment exacerbation was analysed using a Cox proportional hazards model with terms for treatment, reversibility status and percent predicted FEV1 at screening. Exacerbation of COPD is defined by a worsening of symptoms requiring additional treatment. Moderate COPD exacerbation is worsening symptoms of COPD that require treatment with antibiotics and/or systemic corticosteroids. Severe COPD exacerbation is worsening symptoms of COPD that require treatment with in-patient hospitalization. The number of participants with On-Treatment moderate or severe COPD exacerbations are presented.
Time Frame: From the start of double blind study medication until visit 7 (week 12)/Early withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/VI 100/25 µg QD | VI 25 µg QD
Number analyzed (Participants) | 806 | 814
Participants | 69 | 114
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD vs VI 25 µg QD; Test type: Superiority or Other; p < 0.001, Regression, Cox — Nominal p-value; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.43 to 0.78]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of double-blind (DB) study treatment (Visit 2) through the follow up contact (up to 13 weeks).
Description: On-treatment AE or SAE is defined as an AE with an onset date on or after the start date of DB study medication, but not later than one day after the last dose of DB study medication. AEs are reported for participants of the ITT, comprised of all randomized participants who received at least one dose of study medication during the treatment period
Arm/Group | FF/VI 100/25 µg QD | VI 25 µg QD
Serious Adverse Events (participants affected / at risk) | 27/806 | 35/814
Other Adverse Events (participants affected / at risk) | 72/806 | 64/814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg QD (N=806) | VI 25 µg QD (N=814)
Any event (Respiratory, thoracic and mediastinal disorders) | 10 | 19
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 17
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Any event (Infections and infestations) | 6 | 7
Pneumonia (Infections and infestations) | 2 | 4
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Any event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urethral adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Any event (Cardiac disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Any event (Injury, poisoning and procedural complications) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Any event (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Any event (Eye disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 0
Any event (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Any event (Investigations) | 0 | 2
Blood pressure increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Any event (Reproductive system and breast disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Any event (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Any event (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Any event (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg QD (N=806) | VI 25 µg QD (N=814)
Nasopharyngitis (Infections and infestations) | 49 | 48
Headache (Nervous system disorders) | 29 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.